CLINICAL TRIAL: NCT07289646
Title: Functional Lung Avoidance Planning Guided by Lung Perfusion PET/CT Versus Anatomical Planning for Lung Stereotactic Body Radiotherapy
Acronym: Pegasus 2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC23.0220
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stereotactic Body Radiotherapy; 68Ga-MAA; Lung Cancer (Diagnosis)
Keywords: Stereotactic body radiotherapy; 68Ga-MAA lung perfusion; PET/CT; lung radiotherapy
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: (Active Comparator): A conventional anatomical planning will be performed.
  Interventions: Radiation: Conventional anatomical planning radiotherapy
- Experimental group (Experimental): functional planning will be carried out, respecting the standard constraints especially to the tumor and the anatomical lung volume, but also incorporating "lung functional volume" constraints defined by regional lung function mapping.
  Interventions: Radiation: Functional Lung avoidance planning

INTERVENTIONS:
Radiation: Conventional anatomical planning radiotherapy — Conventional anatomical planning will be performed
  Arms: Control group:
Radiation: Functional Lung avoidance planning — Functional Lung Avoidance guided by lung perfusion PET/CT imaging
  Arms: Experimental group

SUMMARY:
Stereotactic body radiotherapy (SBRT) has an increasing role in the treatment of both primary and secondary lung tumors. However, lung SBRT remains associated with significant radiation induced lung injury (RILI). Indeed, the reported incidence of symptomatic radiation induced lung injury (grade≥2) in the published literature is up to 20%. A current challenge of lung SBRT is therefore to better preserve lung function and to reduce pulmonary toxicity.

During standard lung SBRT planning, dose constraints are defined on the anatomical lung volume. This planning considers the lung as functionally uniform and does not take into account the variability of regional lung function distribution. Functional lung avoidance is an emerging concept in lung radiotherapy (RT). The technique aims at personalizing RT treatment planning to individuals' lung functional distribution, by sparing functional pulmonary areas while prioritizing delivery of high doses to non-functional regions.

68Ga-MAA lung perfusion PET/CT is a novel imaging modality for regional lung function assessment. As compared with conventional lung scintigraphy, lung perfusion PET/CT is inherently a vastly superior technology for image acquisition (higher sensitivity and spatial resolution, greater access to respiratory gated acquisition). A more accurate lung functional mapping improves the possibility of functional lung avoidance planning for SBRT.

The hypothesis is that functional lung avoidance planning guided by 68Ga-MAA perfusion PET/CT, while delivering an optimal dose to the tumor, will reduce the frequency of RILI in patients treated with lung SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years planned to be treated in the radiotherapy department of the participating centers with SBRT for primary or secondary lung tumors will be eligible to participate into the study

Exclusion Criteria:

* Inability to give informed consent
* Patientsunder guardianship or curatorship
* Pregnant or breastfeeding women.
* Contraindications to the radiolabeled product infused for lung perfusion PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
To determine whether a functional planning guided by lung perfusion PET/CT imaging is superior to a conventional anatomical planning with regards to the occurrence of grade 2 or higher lung toxicity during the year following lung SBRT. | At year after baseline
  Occurrence of symptomatic RILI (grade≥2 lung toxicity as assessed using the CTCAE 5.0) during the year following lung SBRT. This evaluation will be performed by a medical oncologist blinded from the allocated arm.

SECONDARY OUTCOMES:
quality of life assessment | Measured at 3, 6, 9, and 12 months after baseline
  Quality of life as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), with scores ranging from 0 to 100; higher scores indicate better quality of life for the global health status and functional scales, and worse symptoms for the symptom scales.
quality of life assessment | Measured at 3, 6, 9 and 12 months after baseline
  Quality of life as assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC29), with scores ranging from 0 to 100; higher scores indicate worse symptom burden.
quality of life assessment | Measured at 3, 6, 9, and 12 months after baseline
  Quality of life as assessed by the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire, with index values ranging from -0.594 to 1.0, where higher scores indicate better health-related quality of life.
Grade 3 or higher RILI | Measured at 3, 6, 9, and 12 months after baseline
  Lung toxicity as assessed using the CTCAE 5.0, RTOG and Late effects in normal tissue-subjective objective management analysis (LENT-SOMA) scales
Local tumor control; | Measured at 3, 6, 9, and 12 months after baseline
  Local tumor control;
Progression-free survival; | Measured at 3, 6, 9, and 12 months after baseline
  Progression-free survival
Overall survival. | at 12 months after baseline
  Overall survival

OTHER OUTCOMES:
Decrease of lung perfusion | at 3 months after baseline
  Lung perfusion PET/CT imaging
Overall survival | at 12 months after baseline
  Grade≥2 lung toxicity during the year following lung SBRT

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Brest, Brest, Finistère
  - Centre de Lutte Contre le Cancer Leon Bérard Lyon, Lyon